CLINICAL TRIAL: NCT01207687
Title: Phase 2 Study of Bevacizumab in Children and Adults With Neurofibromatosis Type 2 and Symptomatic Vestibular Schwannoma
Brief Title: Bevacizumab for Symptomatic Vestibular Schwannoma in Neurofibromatosis Type 2 (NF2)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02987; NCI-2012-02987 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); J1002; NA_00034732 (Other: Johns Hopkins University/Sidney Kimmel Cancer Center); 8248 (Other: CTEP); P30CA006973 (NIH); NCT01204463 (obsolete NCT alias)
Record Dates: First submitted 2010-09-01; First posted 2010-09-23 (Estimated); Results first posted 2017-08-17 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Vestibular Schwannoma; Neurofibromatosis Type 2
MeSH Terms: conditions — Neuroma, Acoustic; Neurofibromatosis 2 | interventions — Bevacizumab

ARMS (1):
- Treatment (bevacizumab) (Experimental): Patients receive bevacizumab IV over 30-90 minutes once every 3 weeks. Courses repeat every 6 weeks for up to 48 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab; Other: laboratory biomarker analysis; Procedure: quality-of-life assessment

INTERVENTIONS:
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Other: laboratory biomarker analysis — Correlative studies
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
People who have neurofibromatosis type 2 (NF2) can have tumors that grow on the auditory nerves and cause hearing loss. These tumors are called vestibular schwannomas (VSs), or acoustic neuromas. People with NF2 can also get schwannomas in other parts of their body, as well as tumors called meningiomas and ependymomas. Because VSs can cause hearing loss, many people with NF2 will have treatment to preserve their hearing. This treatment usually involves surgery. Because surgery has risks and is not able to help everyone with VSs, other methods of treatment are being explored. One area of exploration is looking to see if there is a drug that can be taken that might prevent the VSs from growing larger and causing hearing loss or brainstem compression. This study is exploring whether a drug that is approved by the FDA and is currently used to treat other tumors might also work to treat VSs. Based on people who have taken this drug to treat VSs already, there is some reason to think that it might be helpful to certain people with NF2. People enrolled in this study will receive the drug one time every three weeks for one year by infusion. This study will follow subjects over the course of the year that the person is taking the drug and for six months after the drug is stopped. This study is recruiting people who have NF2 and are currently having symptoms of tinnitus, dizziness, and/or hearing loss from their VSs. If you have NF2 and are currently having symptoms caused by your VSs, you may be eligible to participate.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The primary objective of this study is to determine the activity of bevacizumab for treatment of symptomatic vestibular schwannomas (VS) defined as progressive hearing loss in patients with neurofibromatosis type 2 (NF2) based on objective hearing response.

SECONDARY OJBECTIVES:

I. Determine the safety and tolerability of bevacizumab in this patient population on an every three week dosing schedule of 7.5mg/kg for 12 months of therapy.

II. Assess the rate of radiographic response (>= 20% reduction in volume). III. Determine the growth rate of VS using volumetric MRI analysis in comparison to 1-dimensional and 2-dimensional measurements.

IV. Assess changes in function of the auditory system during bevacizumab treatment.

V. Assess the vascular permeability (Ktrans), relative cerebral blood volume/flow, mean transit time, and mean vessel diameter from perfusion-weighted MRI.

VI. Assess the change in circulating endothelial cells, circulating progenitor cells, and plasma angiogenic proteins in subjects receiving bevacizumab treatment.

VII. Observe the impact of bevacizumab on non-VS tumors in patients with NF2 via whole body MRI.

VIII. Explore hearing related QOL measures throughout treatment. IX. Explore the effect of treatment with bevacizumab on auditory function using distortion product optoacoustic emissions (DPOAE) (to be evaluated at NCI only).

OUTLINE:

Patients receive bevacizumab intravenously (IV) over 30-90 minutes once every 3 weeks. Courses repeat every 6 weeks for up to 48 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a confirmed diagnosis of neurofibromatosis 2 by fulfilling National Institute of Health (NIH) criteria or Manchester criteria, or by detection of a causative mutation in the NF2 gene

  * The NIH criteria (82) includes presence of:

    * Bilateral vestibular schwannomas, OR
    * First-degree relative with NF2 and EITHER unilateral eighth nerve mass OR two of the following: neurofibroma, meningioma, glioma, schwannoma, juvenile posterior subcapsular lenticular opacity
  * The Manchester criteria (101) includes presence of:

    * Bilateral vestibular schwannomas, OR
    * First-degree relative with NF2 and EITHER unilateral eighth nerve mass OR two of the following: neurofibroma, meningioma, glioma, schwannoma, juvenile posterior subcapsular lenticular opacity, OR
    * Unilateral vestibular schwannoma AND any two of: neurofibroma, meningioma, glioma, schwannoma, juvenile posterior subcapsular lenticular opacity, OR
    * Multiple meningiomas (two or more) AND unilateral vestibular schwannoma OR any two of: schwannoma, glioma, neurofibroma, cataract
* Patients must have measurable disease, defined as at least one VS >= 1.5 cm (on longest diameter) as measured by contrast-enhanced cranial MRI scan with fine cuts through the internal auditory canal (3 mm slices, no skip)
* Life expectancy of greater than 6 months
* ECOG performance status (Karnofsky >= 60% or Lansky Score >= 60)
* Patients must have normal organ and marrow function as defined below:
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 150,000/mcL or lower limit of institutional normal
* Total bilirubin =< 2 X institutional upper limit of normal
* AST(SGOT)/ALT(SGPT) =< 2.5 X institutional upper limit of normal
* Patients must have recovered from acute toxicity of prior treatment to grade 1 or less unless otherwise specified
* Patients must have a creatinine clearance or radioisotope GFR >= 60ml/min/1.73 m^2 or a normal serum creatinine based on age described in the table below:

  * Age(years) =< 5: 0.8 mg/dL
  * 5 < age (years) =< 10: 1.0 mg/dL
  * 10 < age (years) =< 15: 1.2 mg/dL
  * Age (years) > 15: 1.5 mg/dL
* Subjects must have a VS not amenable to surgery or have refused surgery due to high risk for permanent complications related to surgery (e.g. damage to lower cranial nerve function, facial palsy, risk for cerebrospinal fluid leak, etc.) as determined by a surgeon with experience in management of NF2 associated VS
* Subjects must have had a discussion of all available treatment options and their risks and benefits of these options including surgery, radiation therapy, observation, other clinical trials and expressed their preference for participation in this trial in the informed consent process
* The effects of bevacizumab on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because anti-angiogenic agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness give written informed consent or assent
* Evidence of active disease, defined as progressive hearing loss (with decrease in word recognition score) related to VS (i.e., not due to prior interventions such as surgery or radiation) documented in the preceding 24 months with a word recognition score of < 90% in the target ear
* Proteinuria (including albuminuria) should be screened for by either urine analysis for urine protein creatinine (UPC) ratio or by urine dipstick; if the UPC ratio is greater than or equal to 0.5 or if urine dipstick shows 2+ proteinuria, 24-hour urine protein should be obtained and the level should be < 1000 mg for patient enrollment

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients with nervous system tumors associated with NF2 (e.g., schwannomas, meningiomas, ependymomas, or gliomas) will not be excluded from this clinical trial as long as these tumors do not require treatment with radiation, surgery, or medical treatment at the time of enrollment on trial
* Patients with known hypersensitivity of Chinese hamster ovary cell products, other recombinant human antibodies, or compounds of similar chemical or biologic composition to bevacizumab
* Inability to tolerate periodic MRI scans or gadolinium contrast without general anesthesia
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements
* Clinically significant cardiovascular disease, such as:

  * Inadequately controlled HTN (adult subjects: SBP > 160 mmHg and/or DBP > 90 mmHg despite antihypertensive medication, pediatric subjects: Requirement for antihypertensive treatment prior to enrollment, or diastolic blood pressure > 95th percentile for age)
  * History of CVA within 12 months
  * Myocardial infarction or unstable angina within 12 months
  * New York heart association grade II or greater congestive heart failure
  * Serious and inadequately controlled cardiac arrhythmia
  * Significant vascular disease (e.g. aortic aneurysm, history of aortic dissection)
  * Clinically significant peripheral vascular disease
* Pregnant women (positive pregnancy test) are excluded from this study because bevacizumab is an anti-angiogenic agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with bevacizumab, breastfeeding should be discontinued if the mother is treated with bevacizumab; both fertile men and women must agree to use adequate contraceptive measures during study therapy and for at least 6 months after the completion of bevacizumab therapy; abstinence is considered an adequate contraceptive measure

  * In the event that a minor (age 12-17) who undergoes a pregnancy test as part of the screening process receives a positive result, they will be excluded from the study and their parent(s) of record will be notified of this result
* HIV-positive patients or cancer survivors are eligible for this study if they fulfill all other eligibility criteria
* Inability to perform volumetric measurement of target VS (e.g., due to the MRI artifact from auditory brainstem implant or due to presence of collision tumor (two or more tumors abutting each other) in the cerebellopontine angle); Note: questions about the ability to perform volumetric analysis on a baseline MRI scan should be directed to the study radiologist, Dr. Gregory Sorensen
* Concurrent use of anti-coagulant drugs (not including prophylactic doses), history of coagulopathy, or evidence of bleeding diathesis or coagulopathy
* Imaging (CT or MRI) evidence of newly identified hemorrhage (new within the last in the 6 months prior to enrollment), any history of symptomatic intracranial hemorrhage, or any history of spontaneous intracranial hemorrhage
* Serious or non-healing wound, ulcer or bone fracture
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months prior to day 1
* Invasive procedures defined as follows:

  * Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to Day 1 therapy
  * Brain biopsy within 28 days prior to day 1 of therapy (wounds must be fully healed from brain biopsies performed more than 28 days prior to day 1 of therapy)
  * Anticipation of need for major surgical procedures during the course of the study
  * Core biopsy within 7 days prior to D1 therapy
* Prior treatment with bevacizumab or other VEGF targeting therapies
* Personal history of autoimmune coagulopathy, including idiopathic thrombocytopenia purpura (ITP)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-10; Primary Completion 2013-02 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaishri Blakeley, Principal Investigator — Johns Hopkins University/Sidney Kimmel Cancer Center
Locations (3):
- United States (3):
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - National Cancer Institute, Rockville, Maryland
  - Massachusetts General Hospital, Charlestown, Massachusetts

IPD SHARING:
Plan to Share IPD: No
No individual patient data will be shared

REFERENCES:
- [Result] Blakeley JO, Ye X, Duda DG, Halpin CF, Bergner AL, Muzikansky A, Merker VL, Gerstner ER, Fayad LM, Ahlawat S, Jacobs MA, Jain RK, Zalewski C, Dombi E, Widemann BC, Plotkin SR. Efficacy and Biomarker Study of Bevacizumab for Hearing Loss Resulting From Neurofibromatosis Type 2-Associated Vestibular Schwannomas. J Clin Oncol. 2016 May 10;34(14):1669-75. doi: 10.1200/JCO.2015.64.3817. Epub 2016 Mar 14. PMID 26976425

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Bevacizumab) - All Participants: Bevacizumab IV over 30-90 minutes once every 3 weeks. Courses repeat every 6 weeks for up to 48 weeks in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Bevacizumab) - All Participants
Started | 14
Completed | 12
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Bevacizumab): People with NF2, not eligible for surgery with progressive vestibular schwannoma
Arm/Group | Treatment (Bevacizumab)
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 11
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 30.5 [14 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14
Karnofsky performance status scale [Median (Full Range); unit: units on a scale] — The Karnofsky performance status (KPS) scale is a provider reported measure of functional status. Decile scores are assigned, ranging from 0 to 100. A lower score (minimum 0) represents greater functional impairment. A higher score (maximum 100) represents less functional impairment. KPS can be used measure changes in a patient's functional status.
  units on a scale | 80 [70 to 90]
word recognition score of target ear [Median (Full Range); unit: units on a scale] — The word recognition score (WRS) is the percentage of phonetically-balanced, monosyllabic words that a patient can accurately repeat presented at either most comfortable level or most intelligible level
  units on a scale | 60.5 [13 to 82]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Hearing Response
Description: A hearing response was defined as increased word recognition score above the 95% critical threshold that is maintained across two sequential evaluation time points. The word recognition score (WRS) is the percentage of phonetically-balanced, monosyllabic words that a patient can accurately repeat presented at either most comfortable level or most intelligible level.The proportion of patients with hearing response in the target ear was estimated using a binomial distribution along with 95% confidence intervals.
Time Frame: Baseline to 12 months
Population: All people who underwent treatment were analyzed. Two patients stopped treatment early. One due to toxicity at week 25 and one due to need for medical care not permitted while on treatment at week 49.
Measure: Number (95% Confidence Interval); unit: Proportion with hearing response
Groups:
- Treatment (Bevacizumab) - All Participants: Patients who met all eligibility criteria underwent baseline evaluation and then received bevacizumab 7.5mg/kg IV once every 3 weeks for up to 48 weeks in the absence of disease progression or unacceptable toxicity. Hearing evaluation for word recognition score was evaluated every 12 weeks. Hearing response was defined as improvement beyond the 95% CI maintained across 2 timepoints.
- Treatment (Bevacizumab) - Pediatric Participants Only: All enrolled patients < 18 years of age received bevacizumab 7.5mg/kg IV once every 3 weeks for 12 months.
Arm/Group | Treatment (Bevacizumab) - All Participants | Treatment (Bevacizumab) - Pediatric Participants Only
Number analyzed (Participants) | 14 | 2
Proportion with hearing response | 0.36 [0.13 to 0.65] | 0.50 [0.01 to 0.99]

2. Secondary Outcome: Incidence of Serious or Life Threatening Toxicities
Description: The number of patients with serious or life threatening toxicities (CTCAE grade 3 or above)
Time Frame: Up to 6 months post-treatment
Population: Participants evaluated for serious or life threatening toxicities
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (Bevacizumab) - All Participants: All enrolled patients received bevacizumab 7.5mg/kg IV once every 3 weeks for 12 months.
- Treatment (Bevacizumab) - Pediatric Participants: All enrolled patients < 18 years of age received bevacizumab 7.5mg/kg IV once every 3 weeks for 12 months.
Arm/Group | Treatment (Bevacizumab) - All Participants | Treatment (Bevacizumab) - Pediatric Participants
Number analyzed (Participants) | 14 | 2
Participants | 2 | 0

3. Secondary Outcome: Radiographic Response
Description: The proportion of participants with radiographic response as measured by a >/= 20% reduction in tumor volume from baseline on MRI imaging will be estimated using a binomial distribution.
Time Frame: Baseline to 6 months post-treatment
Measure: Number (95% Confidence Interval); unit: participants
Groups:
- Treatment (Bevacizumab) - All Participants: All enrolled participants received bevacizumab 7.5mg/kg IV once every 3 weeks for up to 12 months.
Arm/Group | Treatment (Bevacizumab) - All Participants | Treatment (Bevacizumab) - Pediatric Participants
Number analyzed (Participants) | 14 | 2
participants | 0.43 [0.18 to 0.71] | 0.50 [0.13 to 0.99]

4. Secondary Outcome: Median Percent Change in Target Vestibular Schwannoma Volume Using Volumetric MRI
Description: The median percent change in the volume of the target vestibular schwannoma using volumetric MRI
Time Frame: Baseline to 12 months
Measure: Median (Full Range); unit: percentage of change in tumor volume
Arm/Group | Treatment (Bevacizumab) - All Participants | Treatment (Bevacizumab) - Pediatric Participants
Number analyzed (Participants) | 14 | 2
percentage of change in tumor volume | 0.5 [-29 to 41] | 10.8 [3.4 to 18.2]

5. Secondary Outcome: Number of Participants With Changes in Function of the Auditory System
Description: The primary distortion product optoacoustic emissions (DPOAE) measurement will be treated non-parametrically (present or absent across time) DPOAE's will be considered present at the frequency of F2 when the distortion product is 6dB above the noise floor. Variables will be analyzed for differences using t-tests if the effects and sample sizes warrant, but this may not be advisable given the small numbers to be accrued.
Time Frame: Baseline to 6 months post-treatment
Population: Distortion product optoacoustic emissions (DPOEs) were only obtained for participants at the NCI site; thus, data from 5 participants were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Bevacizumab) - All Participants
Number analyzed (Participants) | 5
Participants
  Present | 3
  Absent | 2

6. Secondary Outcome: Percent Change in Median Vascular Permeability (Ktrans)
Description: Correlation assessment were planned for imaging parameters and hearing response based on the estimated changes in Ktrans: a MRI measure of vascular permeability. Only 1/14 participants had complete Ktrans data that was amenable to analysis at baseline and week 72. Hence, these statistical analyses were not possible.
Time Frame: Baseline to week 72
Measure: Number; unit: percent change in median Ktrans
Arm/Group | Treatment (Bevacizumab) - All Participants
Number analyzed (Participants) | 1
percent change in median Ktrans | -20

7. Secondary Outcome: Quality of Life Assessed Using Health Survey Short Form-36 (SF-36) - Total Score
Description: The SF-36 is a patient reported outcome. SF-36 (v.1) was administered and was scored according to instructions found on the RAND website. The range of scores is 0 - 100, with a higher value indicating a more favorable health state. The total score is the median of the all the individual items.
Time Frame: Baseline
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment (Bevacizumab) - All Participants
Number analyzed (Participants) | 14
units on a scale | 77.85 [27.36 to 98.19]

8. Secondary Outcome: Quality of Life Assessed Using Health Survey Short Form-36 (SF-36) - Component Scores
Description: The SF-36 is a patient reported outcome. SF-36 (v.1) was administered and was scored according to instructions found on the RAND website. The range of scores is 0 - 100, with a higher value indicating a more favorable health state. Scores are commonly reported as a physical component summary (PCS) and mental component summary (MCS). The PCS and MCS score have been transformed to the T-score metric, which has a mean of 50 and a standard deviation of 10 for the U.S. general population.
Time Frame: Baseline
Measure: Median (Full Range); unit: T-score
Arm/Group | Treatment (Bevacizumab) - All Participants
Number analyzed (Participants) | 14
T-score
  Physical Component Summary (PCS) | 50.67 [22.80 to 61.05]
  Mental Component Summary | 50.79 [33.01 to 56.58]

9. Secondary Outcome: Quality of Life Assessed Using Health Survey Short Form-36 (SF-36) - Total Score
Description: The SF-36 is a patient reported outcome. SF-36 (v.1) was administered and was scored according to instructions found on the RAND website. The range of scores is 1 - 100, with a higher value indicating a more favorable health state. The total score is the median of the all the individual items.
Time Frame: 6 months
Population: One participant was off study at this point secondary to an adverse event and did not complete the questionnaire. Hence, data from 13 of the 14 participants were available for analysis at this time point.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment (Bevacizumab) - All Participants
Number analyzed (Participants) | 13
units on a scale | 80.56 [26.25 to 95.97]

10. Secondary Outcome: Quality of Life Assessed Using Health Survey Short Form-36 (SF-36) - Component Scores
Description: as for outcome 8
Time Frame: 6 months
Population: as for outcome 9
Measure: Median (Full Range); unit: T-score
Arm/Group | Treatment (Bevacizumab) - All Participants
Number analyzed (Participants) | 13
T-score
  Physical Component Score (PCS) | 52.23 [22.73 to 60.45]
  Mental component Summary (MCS) | 54.30 [36.22 to 59.22]

11. Secondary Outcome: Quality of Life Assessed Using Health Survey Short Form-36 (SF-36) - Total Score
Description: as for outcome 7
Time Frame: 12 months
Population: as for outcome 9
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment (Bevacizumab) - All Participants
Number analyzed (Participants) | 13
units on a scale | 75.97 [35.42 to 95.42]

12. Secondary Outcome: Quality of Life Assessed Using Health Survey Short Form-36 (SF-36) - Component Scores
Description: as for outcome 8
Time Frame: 12 months
Population: as for outcome 9
Measure: Median (Full Range); unit: T-score
Arm/Group | Treatment (Bevacizumab) - All Participants
Number analyzed (Participants) | 13
T-score
  Physical Component Summary (PCS) | 47.88 [19.98 to 62.34]
  Mental Component Summary (MCS) | 56.62 [21.10 to 60.94]

13. Secondary Outcome: Quality of Life Assessed Using Health Survey Short Form-36 (SF-36) - Total Score
Description: as for outcome 7
Time Frame: 18 months
Population: One participant had withdrawn consent from the study and did not complete the questionnaire. Hence, data from 13 of the 14 participants were available for analysis at this time point.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment (Bevacizumab) - All Participants
Number analyzed (Participants) | 13
units on a scale | 75.28 [51.67 to 92.64]

14. Secondary Outcome: Quality of Life Assessed Using Health Survey Short Form-36 (SF-36) - Component Scores
Description: as for outcome 8
Time Frame: 18 months
Population: as for outcome 13
Measure: Median (Full Range); unit: T-score
Arm/Group | Treatment (Bevacizumab) - All Participants
Number analyzed (Participants) | 13
T-score
  Physical Component Summary (PCS) | 51.73 [21.07 to 60.02]
  Mental Component Summary (MCS) | 51.51 [26.94 to 67.78]

15. Secondary Outcome: Quality of Life as Assessed by the Speech and Spatial Qualities Questionnaire (SSQ)
Description: The SSQ is a 49 item patient-reported outcome with three subscales: speech understanding (14 questions), spatial location of sounds (17 questions), and the qualities of sounds (18 questions) as they appear to the patient with hearing impairment. Each response is recorded on an 11 point scale (0 - 10), with the anchor points "not at all" (= 0) and "perfectly" (=10). A higher score indicates better hearing. The median score is reported for each subscale. The minimum and maximum scores for the median of each subscale would be 0 and 10, respectively.
Time Frame: baseline
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment (Bevacizumab) - All Participants
Number analyzed (Participants) | 14
units on a scale
  Speech Understanding | 3.2 [0.9 to 6.9]
  Spatial Location of Sounds | 3.2 [0.3 to 8.6]
  Qualities of Sounds | 4.7 [3.1 to 8.9]

16. Secondary Outcome: Quality of Life as Assessed by the Speech and Spatial Qualities Questionnaire (SSQ)
Description: The SSQ is a 49 item patient-reported outcome with three subscales: speech understanding (14 questions), spatial location of sounds (17 questions), and the qualities of sounds (18 questions) as they appear to the patient with hearing impairment. Responses are recorded on a scale from 0 - 10, with the anchor points "not at all" (= 0) and "perfectly" (=10). A higher score indicates better hearing. The median score for each subscale is reported. The minimum and maximum scores for the median of each subscale would be 0 and 10, respectively.
Time Frame: 6 months
Population: At this time point, one participant was off study due to adverse events and did not complete the questionnaire. Three participants did not complete the questionnaire at this time point. Hence, data from 10 participants were available for analysis.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment (Bevacizumab) - All Participants
Number analyzed (Participants) | 10
units on a scale
  Speech Understanding | 4.2 [1.3 to 6.8]
  Spatial Location of Sounds | 4.0 [0.9 to 7.2]
  Qualities of Sounds | 6.8 [3.1 to 8.2]

17. Secondary Outcome: Quality of Life as Assessed by the Speech and Spatial Qualities Questionnaire (SSQ)
Description: as for outcome 16
Time Frame: 12 months
Population: At this time point, one participant was off study due to an adverse event and did not complete the questionnaire. Hence, data from 13 of the 14 participants were available for analysis at this time point.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment (Bevacizumab) - All Participants
Number analyzed (Participants) | 13
units on a scale
  Speech Understanding | 5.4 [2.9 to 8.1]
  Spatial Location of Sounds | 4.8 [1.6 to 9.4]
  Qualities of Sounds | 6.9 [3.1 to 9.7]

18. Secondary Outcome: Quality of Life as Assessed by the Speech and Spatial Qualities Questionnaire (SSQ)
Description: as for outcome 16
Time Frame: 18 months
Population: as for outcome 13
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment (Bevacizumab) - All Participants
Number analyzed (Participants) | 13
units on a scale
  Speech Understanding | 4.1 [2.1 to 7.4]
  Spatial Location of Sounds | 3.6 [0.2 to 9.4]
  Qualities of Sounds | 6.3 [3.2 to 9.6]

19. Secondary Outcome: Quality of Life Assessed by the Tinnitus Reaction Questionnaire (TRQ)
Description: The TRQ is a 26 item patient reported outcome. It is scored using a 5 point Likert scale (0-4). The responses are summed, resulting in a range of 0 - 104 with higher scores indicating more distress related to tinnitus.
Time Frame: baseline
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment (Bevacizumab) - All Participants
Number analyzed (Participants) | 14
units on a scale | 18 [0 to 81]

20. Secondary Outcome: Quality of Life Assessed by the Tinnitus Reaction Questionnaire (TRQ)
Description: as for outcome 19
Time Frame: 6 months
Population: At this time point, one participant was off study due to an adverse event and did not complete the questionnaire. One participant did not complete this questionnaire at this time point. Hence, data from 12 of the 14 participants were available for analysis at this time point.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment (Bevacizumab) - All Participants
Number analyzed (Participants) | 12
units on a scale | 18 [0 to 43]

21. Secondary Outcome: Quality of Life Assessed by the Tinnitus Reaction Questionnaire (TRQ)
Description: as for outcome 19
Time Frame: 12 months
Population: as for outcome 17
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment (Bevacizumab) - All Participants
Number analyzed (Participants) | 13
units on a scale | 10 [0 to 56]

22. Secondary Outcome: Quality of Life Assessed by the Tinnitus Reaction Questionnaire (TRQ)
Description: as for outcome 19
Time Frame: 18 months
Population: At this time point, one participant had withdrawn consent from the study and did not complete the questionnaire. Hence, data from 13 of the 14 participants were available for analysis at this time point.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment (Bevacizumab) - All Participants
Number analyzed (Participants) | 13
units on a scale | 23 [0 to 40]

ADVERSE EVENTS:
Time Frame: From first dose until 6 months off of drug or until resolution of all SAE to baseline, assessed up to 12 months
Description: definition is that used in clinicaltrials.gov
Arm/Group | Treatment (Bevacizumab) - All Participants | Treatment (Bevacizumab) - Pediatric Participants
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/2
Serious Adverse Events (participants affected / at risk) | 2/14 | 0/2
Other Adverse Events (participants affected / at risk) | 13/14 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Bevacizumab) - All Participants (N=14) | Treatment (Bevacizumab) - Pediatric Participants (N=2)
Hypertension (Vascular disorders) | 1 (2) | 0 (0)
Idiopathic thrombocytopenia purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Treatment (Bevacizumab) - All Participants (N=14) | Treatment (Bevacizumab) - Pediatric Participants (N=2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0
ALT increased (Investigations) | 5 (8) | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0
Anorexia (Metabolism and nutrition disorders) | 1 (2) | 0
AST increase (Investigations) | 4 (8) | 0
Bruising (Injury, poisoning and procedural complications) | 2 (2) | 0
CPK increase (Investigations) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Electrocardiogram with prolonged QTc (Investigations) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 1 (1)
Fatigue (General disorders) | 9 (13) | 1 (2)
Headache (Nervous system disorders) | 1 (2) | 1 (2)
Hemoglobinuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 2 (2) | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (4) | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (3) | 1 (2)
Hypomagnesemia (Vascular disorders) | 1 (1) | 0
Increased blood bicarbonate (Investigations) | 1 (1) | 0
Irregular menstruation (Reproductive system and breast disorders) | 2/7 (6) | 1 (4)
Menorrhagia (Reproductive system and breast disorders) | 1/7 (3) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0
Nausea (Gastrointestinal disorders) | 4 (7) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 2 (2) | 0
Oral pain (Gastrointestinal disorders) | 1 (1) | 0
Palpitations (Cardiac disorders) | 2 (2) | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0
Platelet count decreased (Investigations) | 1 (2) | 1 (2)
Proteinuria (Renal and urinary disorders) | 2 (10) | 1 (6)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0
Nasal septum perforation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Vomiting (Gastrointestinal disorders) | 1 (1) | 0
Weight gain (Investigations) | 1 (1) | 0
Weight loss (Gastrointestinal disorders) | 1 (1) | 0
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less